CLINICAL TRIAL: NCT07031050
Title: Robotic Sacrocolpopexy and Sacrocervicopexy - an Observational Study to Confirm the Peri- and Postoperative Safety and Clinical Performance
Acronym: SPARO
Status: Recruiting | Type: Observational
Sponsor: Distalmotion SA (Industry)
Collaborators: Confinis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-03
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Sacrocolpopexy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sacrocolpopexy or sacrocervicopexy — Robotic-assisted sacrocolpopexy or sacrocervicopexy with the Dexter robotic surgery system

SUMMARY:
This study aims to confirm the perioperative and early postoperative safety and clinical performance (efficacy) of the Dexter Robotic System, in patients undergoing robotic-assisted sacrocolpopexy or sacrocervicopexy.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years
* Women with symptomatic stage I or greater pelvic organ prolapse (POP-Q)
* Patient agrees to perform the 6-week follow-up assessment as per Standard of Care

Exclusion Criteria:

* Any planned non-urogynaecological concomitant procedures
* History of previous POP surgery, with the exception of transvaginal approaches without mesh implantation
* Previous surgery and/or radiation for urologic, gastrointestinal or gynecologic cancer
* History of Crohn's disease
* Chronic colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing a sacrocolpopexy or sacrocervicopexy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety outcome | up to 42 days after surgery
  Occurrence of Clavien-Dindo grades III-V adverse events
Primary efficacy outcome | Intraoperative
  Successful completion of the Dexter-assisted procedure, i.e. free of any conversion to an open or fully laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Krankenhaus St. Elisabeth, Damme
  - Universitätsmedizin Essen, Essen
- Switzerland (2):
  - Inselspital Bern, Bern
  - Spitäler FMI AG, Interlaken